CLINICAL TRIAL: NCT02327845
Title: Phenotype, Genotype & Biomarkers in ALS and Related Disorders
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH); St. Jude Children's Research Hospital (Other); ALS Association (Other)
Responsible Party: Principal Investigator, Michael Benatar, Chief of the Neuromuscular Division, Professor of Neurology, University of Miami
Other Study IDs: 20160603; U54NS092091 (NIH)
Record Dates: First submitted 2014-12-24; First posted 2014-12-30 (Estimated); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Amyotrophic Lateral Sclerosis; Frontotemporal Dementia; Primary Lateral Sclerosis; Hereditary Spastic Paraplegia; Progressive Muscular Atrophy; Multisystem Proteinopathy
Keywords: natural history, biomarkers, phenotype, genotype
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Frontotemporal Dementia; Motor Neuron Disease; Spastic Paraplegia, Hereditary; Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, serum, urine and CSF
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Affected: Affected with any of the diseases that are the focus of study by the CReATe Consortium, including ALS, ALS-FTD, HSP, PLS, PMA and MSP.
- Unaffected: Unaffected family members of enrolled affected individuals.

SUMMARY:
The goals of this study are: (1) to better understand the relationship between the phenotype and genotype of amyotrophic lateral sclerosis (ALS) and related diseases, including primary lateral sclerosis (PLS), hereditary spastic paraplegia (HSP), progressive muscular atrophy (PMA), and frontotemporal dementia (FTD); and (2) to develop biomarkers that might be useful in aiding therapy development for this group of disorders.

DETAILED DESCRIPTION:
This study will recruit patients with ALS, ALS-FTD, PLS, HSP, and PMA, with a focus on incident cases. Patients with both familial and sporadic forms of these diseases will be enrolled and followed longitudinally using a standardized set of evaluations. Biological samples (blood, urine, CSF) will be collected from all study participants, and will be used for biomarker discovery and validation. Family members of affected individuals may also be enrolled and asked to contribute DNA and biological samples to aid genetic and biomarker discovery.

ELIGIBILITY:
Inclusion Criteria:

* Member of at least one of the following categories:

  1. Individuals with a clinical diagnosis of ALS or a related disorder, including FTD, HSP, PLS, PMA and MSP (sporadic or familial).
  2. Family member of an enrolled affected individual.
* Able and willing to comply with relevant procedures.

Exclusion Criteria:

* Affected with end or late stage disease.
* A condition or situation which, in the PI's opinion, could confound the study finding or may interfere significantly with the individual's participation and compliance with the study protocol. This includes (but is not limited to) neurological, psychological and/or medical conditions.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with ALS or a related neurodegenerative disorder, including FTD, HSP, PLS, PMA and MSP. Select family members of affected participants.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2015-04; Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Phenotypic correlates of genotype | 24 months
  Using longitudinally collected deep phenotypic data, this project aims to define the natural history (i.e. temporal rate of disease progression) of the motor and frontotemporal system (behavior, cognition and language) phenotypes of ALS and related disorders in patients with identifiable genetic mutations.
Genetic determinants of phenotype | 24 months
  By combining longitudinally collected deep phenotypic data with deep genetic data (e.g. whole exome or whole genome sequencing), this project aims to define genetic variants that are associated with identifiable phenotypic features in patients with ALS and related disorders.

OTHER OUTCOMES:
Biomarkers | 24 months
  Biomarkers relevant to therapeutic development

CONTACTS AND LOCATIONS:
Overall Officials: Michael Benatar, DPhil, Principal Investigator — University of Miami
Locations (15):
- United States (13):
  - Stanford University, Palo Alto, California
  - University of California San Diego (UCSD), San Diego, California
  - California Pacific Medical Center (CPMC), San Francisco, California
  - University of Miami, Miami, Florida
  - University of Iowa, Iowa City, Iowa
  - Kansas University Medical Center (KUMC), Kansas City, Kansas
  - Twin Cities ALS Research Consortium, Minneapolis, Minnesota
  - Wake Forest University, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Southwestern (UTSW), Dallas, Texas
  - University of Texas Health Science Center San Antonio (UTHSCSA), San Antonio, Texas
  - University of Virginia (UVA), Charlottesville, Virginia
- Eberhard Karls University of Tübingen, Tübingen, Germany
- University of Cape Town, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Benatar M, Macklin EA, Malaspina A, Rogers ML, Hornstein E, Lombardi V, Renfrey D, Shepheard S, Magen I, Cohen Y, Granit V, Statland JM, Heckmann JM, Rademakers R, McHutchison CA, Petrucelli L, McMillan CT, Wuu J; CReATe Consortium PGB1 Study Investigators. Prognostic clinical and biological markers for amyotrophic lateral sclerosis disease progression: validation and implications for clinical trial design and analysis. EBioMedicine. 2024 Oct;108:105323. doi: 10.1016/j.ebiom.2024.105323. Epub 2024 Sep 12. PMID 39270623
- [Derived] Benatar M, Macklin EA, Malaspina A, Rogers ML, Hornstein E, Lombardi V, Renfrey D, Shepheard S, Magen I, Cohen Y, Granit V, Statland JM, Heckmann JM, Rademakers R, McHutchison CA, Petrucelli L, McMillan CT, Wuu J. Prognostic Clinical and Biological Markers for Amyotrophic Lateral Sclerosis Disease Progression: Validation and Implications for Clinical Trial Design and Analysis. medRxiv [Preprint]. 2024 Aug 13:2024.08.12.24311876. doi: 10.1101/2024.08.12.24311876. PMID 39185513